CLINICAL TRIAL: NCT04582578
Title: Resynchronization for Ambulatory Heart Failure Trial in Patients With Preserved LV Function (RAFT-Preserved)
Brief Title: Resynchronization for Ambulatory Heart Failure Trial in Patients With Preserved LV Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Anthony Tang (Other)
Responsible Party: Sponsor-Investigator, Anthony Tang, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO 3310
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: LBBB; Medical Therapy; Sinus Rhythm; Preserved LV Function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a multi-centre randomized controlled trial with a prospective randomized open blinded endpoint trial (PROBE) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will be treated with practice guideline optimal medical therapy for HF.
- BiV-CRT (Experimental): The experimental group will be treated with CRT in addition to optimal medical therapy for HF. In addition, the trial will further compare two methods of delivering CRT. One experimental group will receive BiV-CRT, while the second experimental group will receive Conduction System(CS)-CRT.
  Interventions: Device: CRT
- CS-CRT (Experimental): The experimental group will be treated with CRT in addition to optimal medical therapy for HF. In addition, the trial will further compare two methods of delivering CRT. One experimental group will receive BiV-CRT, while the second experimental group will receive Conduction System(CS)-CRT.
  Interventions: Device: CRT

INTERVENTIONS:
Device: CRT — The experimental group will be treated with CRT in addition to optimal medical therapy for HF. In addition, the trial will further compare two methods of delivering CRT. One experimental group will receive BiV-CRT, while the second experimental group will receive CS-CRT
  Arms: BiV-CRT; CS-CRT

SUMMARY:
This trial will compare two management strategies for HF patients with preserved LV function in sinus rhythm and LBBB. The control group will be treated with practice guideline optimal medical therapy for HF. The experimental group will be treated with CRT in addition to optimal medical therapy for HF. In addition, the trial will further compare two methods of delivering CRT. One experimental group will receive BiV-CRT, while the second experimental group will receive CS-CRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA class II-IVa HF symptoms and are on diuretic therapy
* LVEF > 35% (stratify by LVEF 36-49% and LVEF ≥ 50%), and recovered LVEF (previously LVEF ≤ 35%, but improved to LVEF > 35% with medical therapy)
* Patients with LVEF ≥ 50% must also have either left atrial enlargement (any of the following: LA diameter ≥3.8 cm, LA length ≥5.0 cm, LA volume ≥55 ml, LA volume index (LAVi) ≥29 mL/m2) or LV hypertrophy (LV mass index (LVMI) ≥115 g/m2 for males and ≥ 95g/m2 for females)
* LBBB and QRS duration ≥ 140 msec. for men or ≥ 130 msec. for women, and with mid-QRS notching or slurring in ≥ 2 leads
* Patients may have permanent RV pacing with a QRS duration ≥180ms
* Patients may have permanent atrial fibrillation with good rate control defined as a resting heart rate of ≤80 bpm at rest and ≤110 bpm with 6-minute walk test
* NT-proBNP ≥ 600 pg/ml on stable medical therapy without previous heart failure hospitalization in the last 12 months, or ≥400 pg/ml on stable medical therapy if there was a heart failure hospitalization within the previous 12 months
* Appropriate pharmacological treatment of HF and co-morbidities.
* Stable diuretic and other HF medications for at least four weeks

Exclusion Criteria:

* Serum creatinine >180 μmol/L; or estimated glomerular filtration rate [eGFR] ≤30 mL/min/1.73 m2, calculated using the Modification of Diet in Renal Disease formula
* In-hospital patients with acute cardiac or non-cardiac illness that requires intensive care
* Acute coronary syndrome (including MI) <4 weeks
* Coronary revascularization (CABG or PCI) < 3 months
* Uncorrected or uncorrectable primary valvular disease
* TAVI < 3 months
* Restrictive, or reversible form of cardiomyopathy, cardiac amyloidosis
* Severe primary pulmonary disease such as cor pulmonale, primary pulmonary hypertension (may include secondary pulmonary hypertension, if mean pulmonary pressure is ≤ 70 mm Hg)
* Expected to undergo cardiac transplantation within one year (status I)
* Patients with a life expectancy of less than one year from non-cardiac cause.
* Patients included in other clinical trials that will affect the objectives of this study
* Patients who are pregnant/intend to get pregnant
* Those unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
NTproBNP measurement | 6 Months
  The co-primary outcome measure is NTproBNP as measured at 6 months.
6-minute walk distance | 6 Months
  The co-primary outcome measure is 6 minute hall walk distance as measured at 6 months.
Quality of Life (QoL) score | 6 Months
  The co-primary outcome measure is quality of life as measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ) score. The MLHFQ consists of 21 questions answered on a 0-5 likert scale, with higher scores indicating a stronger impact of heart failure on QoL.

SECONDARY OUTCOMES:
Ventricular arrhythmia burden determined by the device capture of arrhythmias and adjudication by a device review committee blinded to patient's treatment allocation | 6 Months
  The secondary outcome measure is Ventricular arrhythmia burden determined by the device as measured at 6 months.
LV reverse remodeling (LVESVi on echocardiography) | 6 Months
  The secondary outcome measure is LV reverse remodeling as measured by LVESVi on echocardiography at 6 months.
LVEF | 6 Months
  The secondary outcome measure is LVEF as measured by echocardiography at 6 months.
A composite of all-cause mortality and HF events | 6 Months
  The secondary outcome measure a composite of all-cause mortality and HF events at 6 months.
Packer Composite Clinical Outcome Score | 6 Months
  The secondary outcome measure is Packer Composite Clinical Outcome Score at 6 months. The Packer Clinical Composite Score classifies each patient into 1 of 3 categories (improved, worsened, unchanged), and is determined using clinical outcomes, heart failure status, and patient symptoms. Patients are considered improved if at the final visit they experienced in the patient assessment of a pre-specified scale but did not experience any major adverse clinical events throughout the trial. If considered worse, patients experienced a major clinical event during the planned duration of double-blind treatment or reported worsening at their final visit. And if considered unchanged, patients would be considered neither improved nor worse.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No